CLINICAL TRIAL: NCT04877691
Title: A Multicentre, Randomised, Double-Blind, Placebo-controlled, Phase 3 Study Evaluating the Efficacy and Safety of Subcutaneous Anifrolumab in Adult Patients With Systemic Lupus Erythematosus
Brief Title: Subcutaneous Anifrolumab in Adult Patients With Systemic Lupus Erythematosus
Acronym: Tulip SC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3465C00001; SZA64400; 2020-004529-22 (EudraCT Number)
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosuss Anifrolumab, Adult patients, BICLA, glucocorticoids, Immunosuppressant(s), sub-cutaneous
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double Blind (Participant, Care Provider and Investigator) and OLE
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (Experimental): Solution for injection in aPFS
  Interventions: Drug: Medi-546
- Placebo (Placebo Comparator): Solution for injection in aPFS
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Medi-546 — Patients will have IP administered or will self-administer IP under supervision by site staff at Week 0 and Week 1 and, for patients participating in the OLE period, at Week 52. For weekly doses coinciding with subsequent on-site visits, patients will also have IP administered or will self-administer IP under supervision by site staff, and in addition will receive a set of kits (including back-up kits) for at-home administration.
  Arms: Anifrolumab
Drug: Placebo — Solution for injection in aPFS
  Arms: Placebo

SUMMARY:
The purpose of this study is evaluating the efficacy and safety of SC antifrolumab in adult patients with moderate -to-severe SLE despite receiving standard therapy

DETAILED DESCRIPTION:
This is a Phase 3, multicentre, multinational, randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of a subcutaneous treatment regimen of anifrolumab versus placebo in participants with moderately to severely active, autoantibody-positive systemic lupus erythematosus (SLE) while receiving standard of care (SOC) treatment. Participants must be taking either 1 or any combination of the following: oral glucocorticoids, antimalarial, and/or immunosuppressants. The study will be performed in adult participants of 18 to 70 years of age.

Approximately 360 participants receiving SOC treatment will be randomised in a 1:1 ratio to receive a fixed subcutaneous dose of anifrolumab or placebo administered once weekly via an accessorized prefilled syringe and with the primary endpoint evaluated at Week 52. Subjects who complete Week 52 may enter into open-label extension (OLE). All patients who enter the OLE Period will receive a fixed subcutaneous dose of anifrolumab for up to 52 weeks. Study intervention will be administered SC via an accessorised prefilled syringe (aPFS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a diagnosis of pediatric or adult SLE according to the ACR 1997 revised criteria for ≥ 24 weeks prior to signing the ICF
2. To be eligible a patient must have SLEDAI-2K ≥ 6 points and "Clinical" SLEDAI-2K score ≥4 points at screening
3. BILAG2004 with at least 1 of the following:

   1. BILAG2004 level A disease in ≥ 1 organ system
   2. BILAG2004 level B disease in ≥ 2 organ systems
4. Physician's Global Assessment (PGA) score ≥ 1.0 on a 0 to 3 VAS at Screening
5. Antinuclear antibody, and/or Anti-dsDNA and/oranti-Smith positive at Screening,
6. Must be on stable background standard therapy with DMARD, glucocorticoids or anti-malarials alone or in combinations.

   Exclusion Criteria:
7. Active severe or unstable neuropsychiatric SLE
8. Active severe SLE-driven renal disease
9. History of any non-SLE disease that has required treatment with oral or parenteral corticosteroids for more than a total of 2 weeks within the last 24 weeks prior to signing the ICF.
10. History of recurrent infection requiring hospitalization and IV antibiotics (eg, 3 or more of the same type of infection over the previous 52 weeks).
11. Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the patient to infection, or a positive result for human immunodeficiency virus (HIV) infection confirmed by central laboratory at Screening.
12. At Screening, confirmed positive test for hepatitis B serology and positive test for hepatitis C antibody
13. Any severe case herpes zoster infection at any time prior to Week 0 (Day 1),
14. Opportunistic infection requiring hospitalization or IV antimicrobial treatment within 3 years of randomization.
15. History of cancer, apart from:

    1. Squamous or basal cell carcinoma of the skin treated with documented success of curative therapy ≥ 3 months prior to Week 0 (Day 1)
    2. Cervical cancer in situ treated with apparent success with curative therapy ≥ 1 year prior to Week 0 (Day 1).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) response | At week 52
  BICLA response is a composite binary endpoint whereby responders are defined by meeting all of the following criteria:
  * Improvement from baseline in disease activity as measured by BILAG-2004. Improvement is defined as a reduction of all baseline BILAG-2004 A to B/C/D and baseline BILAG-2004 B to C/D and no BILAG-2004 worsening in other organ systems, where worsening is defined as ≥ 1 new BILAG-2004 A or ≥ 2 new BILAG 2004 B.
  * No worsening from baseline in SLEDAI-2K, where worsening is defined as an increase from baseline of > 0 points in SLEDAI-2K.
  * No worsening from baseline in the patient's lupus disease activity, where worsening is defined as an increase ≥ 0.30 points on a 3-point PGA VAS.

SECONDARY OUTCOMES:
Time to first BICLA response sustained through Week 52 | Baseline through to Week 52
  Time from first dose to first BICLA response that is consecutively maintained through Week 52
BICLA response with maintained low (or reduced) use of oral corticosteroid (OCS) | At week 52
  Response is defined by being a BICLA responder at Week 52 and having maintained low (or reduced) OCS use through Week 52. Maintained OCS use is defined as follows:
  * If baseline OCS ≥ 10 mg/day an OCS dose of ≤ 7.5 mg/day prednisone or equivalent must be achieved by Week 40 and an OCS dose ≤ 7.5 mg/day prednisone or equivalent must be maintained from Week 40 to Week 52.
  * If baseline OCS < 10 mg/day, OCS dose at Week 40 must be less than or equal to OCS dose at baseline, with no increase from Week 40 OCS dose between Week 40 and Week 52.
Time to flare | Baseline through to Week 52
  Flare defined as either 1 or more BILAG 2004 A or 2 or more BILAG 2004 B compared to previous visit
Maintained oral corticosteroid (OCS) reduction among patients with baseline OCS ≥10 mg/day. | At week 52
  Achieving maintained OCS reduction through Week 52 is defined by meeting all of the following criteria:
  * Achieve an OCS dose of ≤ 7.5 mg/day prednisone or equivalent by Week 40
  * Maintain an OCS dose ≤ 7.5 mg/day prednisone or equivalent from Week 40 to Week 52
  * No discontinuation of investigational product
  * No use of restricted medications beyond the protocol allowed threshold before assessment
Annualized flare rate | Baseline through to Week 52
  Flare defined as either 1 or more BILAG 2004 or 2 or more BILAG2004 B compared to previous visit
SRI4 | At week 52
  Proportion of patients achieving a SRI of ≥ 4 (SRI[4]) response at Week 52, defined by meeting all of the following criteria:
  Reduction from baseline of ≥ 4 points in the SLEDAI-2K No new organ systems affected as defined by 1 or more BILAG-2004 A or 2 or more BILAG 2004 B items compared to baseline using BILAG-2004 No worsening from baseline in the patients' lupus disease activity, where worsening is defined by an increase ≥ 0.30 points on a 3-point PGA VAS.

OTHER OUTCOMES:
Adverse Event Overview | Up to 2 years 4 months
  Overview of AEs, SAEs and AESIs

CONTACTS AND LOCATIONS:
Locations (107):
- United States (30):
  - Research Site, Birmingham, Alabama
  - Research Site, Paradise Valley, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, El Cajon, California
  - Research Site, Fullerton, California
  - Research Site, Hemet, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Menifee, California
  - Research Site, Upland, California
  - Research Site, Aurora, Colorado
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Idaho Falls, Idaho
  - Research Site, Flint, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Newark, New Jersey
  - Research Site, Las Cruces, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Potsdam, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Grapevine, Texas
- Argentina (10):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Mendoza
  - Research Site, Pergamino
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, Salta
  - Research Site, San Isidro
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
- Bulgaria (5):
  - Research Site, Kardzhali
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sevlievo
  - Research Site, Sofia
- Chile (3):
  - Research Site, Osorno
  - Research Site, Santiago
  - Research Site, Valdivia
- Colombia (5):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Chía
  - Research Site, Montería
- Germany (4):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Leipzig
  - Research Site, Tübingen
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Székesfehérvár
  - Research Site, Veszprém
- Japan (15):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Hamamatsu
  - Research Site, Hiroshima
  - Research Site, Itabashi-ku
  - Research Site, Kita-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Meguro-ku
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Sagamihara-shi
  - Research Site, Sasebo-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
- Mexico (7):
  - Research Site, Chihuahua City
  - Research Site, Culiacán
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mexicali
  - Research Site, Mérida
  - Research Site, México
- Research Site, Quezon City, Philippines
- Poland (9):
  - Research Site, Katowice
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Nowa Sól
  - Research Site, Ustroń
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
- Thailand (2):
  - Research Site, Muang
  - Research Site, Rachathewi
- Ukraine (4):
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (3):
  - Research Site, Doncaster
  - Research Site, Leeds
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home